CLINICAL TRIAL: NCT01732432
Title: Endometriosis and Frequency of Endometriosis-associated Ovarian Carcinomas (EAOC) - Epidemiological and Molecular Pathological Aspects
Brief Title: Endometriosis and Frequency of Endometriosis-associated Ovarian Carcinomas (EAOC)
Acronym: EAOC
Status: Withdrawn | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 210/12
Record Dates: First submitted 2012-11-18; First posted 2012-11-22 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Endometrioid Carcinoma; Clear Cell Carcinoma; Endometriosis
MeSH Terms: conditions — Carcinoma, Endometrioid; Adenocarcinoma, Clear Cell; Endometriosis

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to determine whether a relationship exists between a previously established diagnosis of endometriosis and the consecutive risk of developing a clear cell or endometrioid ovarian carcinoma. All histopathological records since 1980 with these diagnoses (endometriosis, clear cell and endometrioid ovarian carcinoma) will be reviewed. Cancer registry data will be assessed to investigate differences in survival of women with endometriosis-associated ovarian carcinomas and those ovarian carcinoma patients without previous diagnosis of endometriosis.

ELIGIBILITY:
Inclusion Criteria:

* endometrioid ovarian carcinoma
* clear cell ovarian carcinoma
* endometriosis, atypical endometriosis
* borderline tumors with endometriosis

Exclusion Criteria:

* undifferentiated carcinomas
* germ cell tumors
* sex cord-stromal tumors

Ages: 30 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care hospital, university hospital
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-10; Primary Completion 2013-08 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
incidence and clinical outcome of endometriosis-associated ovarian carcinomas | 30 years

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Obermann, MD, Dr., Principal Investigator — University Hospital Basel, University of Basel; Ellen C Obermann, MD, Principal Investigator — Institute of Pathology, University Hospital Basel, University of Basel